CLINICAL TRIAL: NCT05979883
Title: A Randomized Evaluation of Machine Learning Assisted Radiation Treatment Planning Versus Standard Radiation Treatment Planning
Brief Title: Randomized Evaluation of Machine Learning Assisted Radiation Treatment Planning vs Standard Radiation Treatment Planning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Daniel J. Ma, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMROR2371; 23-004732 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Cancer Head Neck; Cancer, Head; Cancer Neck
Keywords: MLAP (Machine Learning Adaptive Planning); RapidPlan
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm A: Standard of care (SOC) treatment planning (Other): Patients randomized to the SOC treatment planning arm will receive a treatment planning computed tomography (CT) scan followed by dosimetric planning with a medical dosimetrist; and the plan will be reviewed by a medical physicist and radiation oncologist. This is the current standard practice for all radiation oncology patients.
  Interventions: Radiation: Radiation Therapy Standard of Care (SOC)
- Arm B: Machine Learning Assisted Planning (MLAP) (Active Comparator): Patients randomized to the MLAP arm will receive a treatment planning scan followed by MLAP through the RapidPlan module produced by Varian. Of note, RapidPlan is an FDA cleared module with treatment planning being the approved usage for the program. The RapidPlan module has site specific treatment packages for different disease sites. These separate disease specific packages have different capabilities. For example, the Head and Neck package currently audits dosimetrist-generated plans for possible improvements. The MLAP arm of the trial will leverage the RapidPlan module's full capabilities upwards to the FDA-approved usage.
  Interventions: Radiation: Machine Learning Assisted Radiation (MLAP) RapidPlan

INTERVENTIONS:
Radiation: Machine Learning Assisted Radiation (MLAP) RapidPlan — Radiation therapy simulation, target delineation, dosing, localization, and follow-up will be followed per standard of care practices and/or at the discretion of the treating radiation oncologist. To elaborate, patients will receive a treatment planning CT (computed tomography) scan, followed by normal tissue delineation through the physician and/or medical dosimetry assistant, followed by target delineation by the physician, followed by radiation treatment planning with the dosimetrist and medical physicist. The preliminary plan will be run through the RapidPlan module, which will give a list of possible improvements to the plan. The dosimetrist will then make an amendment to the plan according to RapidPlan suggestions, followed by plan change requests and approval by the physician.
  Arms: Arm B: Machine Learning Assisted Planning (MLAP)
Radiation: Radiation Therapy Standard of Care (SOC) — Radiation therapy simulation, target delineation, dosing, localization, and follow-up will be followed per standard of care practices and/or at the discretion of the treating radiation oncologist. To elaborate, patients will receive a treatment planning CT (computed tomography) scan, followed by normal tissue delineation through the physician and/or medical dosimetry assistant, followed by target delineation by the physician, followed by radiation treatment planning with the dosimetrist and medical physicist, followed by plan change requests and approval by the physician.
  Arms: Arm A: Standard of care (SOC) treatment planning

SUMMARY:
The purpose of this study is to determine the magnitude of clinical benefit achieved through machine learning assisted radiation treatment planning (MLAP) on post-treatment clinical outcomes such as acute toxicity and patient reported outcomes.

DETAILED DESCRIPTION:
This is a randomized phase III trial to evaluate the effectiveness of MLAP compared to Standard of Care. Patients will undergo a randomization procedure with a variable allocation ratio where the first third of patients are randomized 3:1 in favor of SOC, the next third randomized 1:1, and the last third randomized 1:3 in favor of MLAP. This is done to give dosimetrists time to optimize the MLAP workflow. Since the treatment team may learn to improve their treatment planning process in the SOC arm through interactions with RapidPlan, as a sensitivity analysis, the primary and secondary goals will be re-analyzed including time of registration as a moderator of the treatment effect.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at time of registration
* Receiving curative intent intensity modulated radiotherapy for head and neck primary cancer at the discretion of the treating medical doctor (MD)
* Provide written informed consent or allow legally authorized representative to consent on behalf of a participant
* Willing to return to enrolling institution for study follow-up visit

Exclusion Criteria:

* Incarcerated
* Unable to provide informed consent
* Prior Head and Neck (H&N) radiation therapy
* Planned radiation dosing LK<30 Gy or >76 Gy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2025-10-29 (Actual); Study Completion 2025-10-29 (Actual)

PRIMARY OUTCOMES:
Change in swallowing score | Baseline (up to 30 days prior to treatment planning); up to 6 months
  Will be assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Head and Neck module (EORTC QLQ-H&N35). The EORTC QLQ-H&N35 is a 35-item questionnaire used to assess symptoms encountered specifically by patients with head and neck cancer. The H&N35 consists of 7 multiple-item scales (Pain, Swallowing, Senses, Speech, Social eating, Social contact, and Sexuality), in addition to 11 single items (e.g., Opening mouth, Sticky saliva, Dry mouth, etc.). Scores are combined into an overall score ranging from 0=Best to 100=Worst. Swallowing score will be measured at baseline (up to 30 days prior to treatment planning), at the end of Radiation Treatment (+ 14 days), and 3 months post Radiation Treatment (+/-30 days from 3 months post-radiotherapy).

SECONDARY OUTCOMES:
Change in physician-reported toxicities | Baseline; up to 6 months
  Assessed according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Toxicities will be recorded at baseline (up to 30 days prior to treatment planning), at the end of Radiation Treatment (+14 days), and 3 months post Radiation Treatment (+/-30 days from 3 months post-radiotherapy).
Difference in treatment plan quality metrics (PQMs) across treatment arms | Baseline; up to 6 months
  Treatment PQM is a continuous-valued function depending on selected dose-volume histogram statistics for 5 organs-at-risk. Comparisons between treatment arms will be made.
Difference in time to complete treatment planning | Baseline; up to 6 months
  Treatment planning time is defined as the time in minutes from the end of physician contouring to the end of physician plan approval.

OTHER OUTCOMES:
Difference in quality of life scores | Baseline; up to 6 months
  Quality of life scores will be compared between arms, as measured by the 6 remaining subscales and 11 single item scores of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Head and Neck module (EORTC QLQ-H&N35). EORTC scores will be recorded at baseline (up to 30 days prior to treatment planning), at the end of Radiation Treatment (+14 days), and 3 months post Radiation Treatment (+/-30 days from 3 months post-radiotherapy).
Change in dose-volume histograms (DVHs) | Baseline; up to 6 months
  DVH statistics will be compared between treatment arms within cohorts of planned radiation dose (30-54 Gy vs. 54-66 Gy vs. 66-76 Gy) and laterality (bilateral vs. unilateral).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. Ma, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (6):
- United States (6):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials